CLINICAL TRIAL: NCT06112028
Title: Clinical Study of Tongxinluo Capsule in Preventing and Treating Restenosis After Intracranial and External Arterial Stenting
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yanbin Li (Other)
Responsible Party: Sponsor-Investigator, Yanbin Li, Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07
Record Dates: First submitted 2023-10-08; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Stent Restenosis
Keywords: traditional Chinese medicine; Stent Restenosis
MeSH Terms: interventions — tongxinluo

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): In addition to oral aspirin enteric coated tablets (0.1g qd), Clopidogrel bisulfate tablets (75mg qd), rosuvastatin calcium tablets (10mg qd) or atorvastatin calcium tablets (20mg qd), Tongxinluo capsule (Shijiazhuang Yilin Pharmaceutical Co., LTD.) was added to 0.78g TID for continuous treatment for 12 months.
  Interventions: Drug: Tongxinluo capsule; Other: Primary therapy
- control group (Sham Comparator): Take aspirin enteric coated tablets (0.1g qd), Clopidogrel bisulfate tablets (75mg qd), Rosuvastatin calcium tablets (10mg qd) or atorvastatin calcium tablets (20mg qd) orally.
  Interventions: Other: Primary therapy

INTERVENTIONS:
Drug: Tongxinluo capsule — On the basis of conventional treatment, the study participants in the experimental group were given Tongxinluo capsule for 12 months.
  Arms: Experimental group
Other: Primary therapy — Routine oral aspirin enteric-coated tablets, clopidogrel bisulfate tablets and rosuvastatin calcium tablets (or atorvastatin calcium tablets)

SUMMARY:
Intrastent restenosis is a common complication after intracranial and extracranial arterial stenting and an important cause of recurrent ischemic stroke. Studies have shown that Tongxinluo capsule can protect the injured inner cells, reduce inflammation, inhibit the proliferation and migration of smooth muscle cells, inhibit the proliferation of plaque and nourish blood vessels, and resist arteriosclerosis. This study was a multicenter prospective randomized controlled clinical trial. Participants with intracranial and extracranial atherosclerotic stenosis who successfully underwent arterial stenting were included in the study, and were divided into Tongxinluo test group and control group. Clinical and related auxiliary examination data were collected at each follow-up point. To explore the effectiveness and potential mechanism of Tongxinluo capsule in preventing and treating restenosis after intracranial and external arterial stenting, and to provide reference for expanding clinical use of traditional Chinese medicine.

DETAILED DESCRIPTION:
Study participants aged 45-80 years who met the criteria for symptomatic or asymptomatic cerebral artery stenosis and successfully underwent cerebrovascular stenting were randomly divided into test group and control group. On the basis of routine oral treatment ,participants in experimental group were given Tongxinluo capsule. The control group received routine oral treatment. The routine follow-up sites were 1, 3, 6 and 12 months, and clinical data and blood were collected at the initial diagnosis and each follow-up site. SPSS software was used to analyze whether Tongxinluo capsule could reduce restenosis after intracranial and extracranial arterial stenting. During the follow-up, the adverse reactions such as bleeding and gastrointestinal tract were observed.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of symptomatic cerebral artery stenosis study participants met the above diagnostic criteria; Participants in the study with asymptomatic cerebral artery stenosis or asymptomatic cerebral artery stenosis met the indications for stent implantation in the Chinese Guidelines for Intravascular Interventional Treatment of Ischemic Cerebrovascular Diseases 2015, and successfully underwent cerebrovascular stenting (residual stenosis after vascular opening ≤30% after stent implantation).

  * I am 45-80 years old and I and my family members agree to participate in this study.

    * It can tolerate statin and platelet therapy without serious complications.

Exclusion Criteria:

* Patients with other intracranial lesions;

  * Recent bleeding history or bleeding tendency;

    * Patients with severe cardiac, liver and renal insufficiency, hypertension and diabetes were not well controlled;

      (4) Severe symptoms of stroke or neurological impairment and unstable symptoms after surgery;

      (5) Severely infected persons who cannot be controlled;

      ⑥ Patients who stop taking medicine for more than 2 months for various reasons;

      ⑦ Taking proprietary Chinese medicine or traditional Chinese medicine with similar efficacy.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Changes of vascular stenosis rate after intracranial and extracranial arterial stenting | The 12th month
  According to NASCET experimental measurement standards, stenosis rate = (normal vascular lumen diameter - residual diameter at stenosis)/normal vascular lumen diameter *100%. Comparison of CTA or DSA to evaluate the change of vascular stenosis rate after intracranial and extracranial arterial stenting; The incidence of cerebral ischemic events and intracranial hemorrhage events (responsible vessels and non-responsible vessels) were assessed by MR. Blood routine, liver and kidney function, blood lipids and hsCRP were recorded. The incidence and mortality of symptomatic intracranial hemorrhage were analyzed. Adverse events (e.g. abdominal pain, diarrhea, nausea, vomiting, bleeding, etc.)